CLINICAL TRIAL: NCT00559026
Title: Phase I/II Clinical Trial for the Evaluation of the Interaction Between Chemotherapy and Immunotherapy in Melanoma Patients
Brief Title: Phase I/II Study of Chemo-Immunotherapy Combination in Melanoma Patients
Acronym: DTIC-melvacc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Collaborators: Regina Elena Cancer Institute (Other); University of Rome Tor Vergata (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISS-DTIC-melvacc1; 2007-006447-42
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Biological: Melan-A
- 2 (Experimental)
  Interventions: Other: Melan-A plus Dacarbazine

INTERVENTIONS:
Biological: Melan-A — i.d. injections of Melan-A: 26-35 (A27L) and gp100: 209-217 (210M) peptides (250 µg each) formulated in Montanide ISA-51 plus s.c. injection of 3MU IFN-α, as an adjuvant on day 1 and 8 every 21 days for a total of 5 courses
  Arms: 1
Other: Melan-A plus Dacarbazine — Dacarbazine plus vaccine: the vaccination schedule as in arm 1 was combined with DTIC (800 mg/mq i.v.) administered one day before each vaccine administration according to the standard treatment.
  Arms: 2

SUMMARY:
This phase I/II study is directed at evaluating safety and immunogenicity of a melanoma peptide vaccine in combination or not with Dacarbazine administration in melanoma patients

DETAILED DESCRIPTION:
Recently, it is becoming increasingly accepted that, in order to induce a clinically effective antitumor response, immunotherapy needs to be combined with chemotherapy. Thus, the traditional perception that chemotherapy and immunotherapy act through unrelated mechanisms which may be antagonistic is challenged on the premises that a selected panel of drugs can induce an immunogenic cell death producing specific danger signals. Furthermore, chemotherapy combined to immunotherapy may affect antigen cross-presentation, induce a "cytokine storm", reduce the number of regulatory T cells and activate homeostatic lymphoid proliferation. Our previous results obtained in a mouse model, demonstrated that drug-induced cytokines can favour antitumor immunity. Based on this observation, we explored whether the administration of dacarbazine (DTIC) in disease-free melanoma patients in combination with peptide vaccination could result into an improved anti tumor immune response.

Patients included in the study were assigned to two treatment arms either receiving anti-tumor vaccination with Melan-A and gp100 analog peptides alone (arm 1) or in combination with DTIC pre-treatment (arm 2).

Arm 1, vaccine alone: patients received i.d. injections of Melan-A: 26-35 (A27L) and gp100: 209-217 (210M) peptides (250 µg each) formulated in Montanide ISA-51 plus s.c. injection of 3MU IFN-α, as an adjuvant on day 1 and 8 every 21 days for a total of 5 courses (10 vaccinations). Both peptides and IFN-α were injected in close but separate sites next to local lymph nodes.

Arm 2, DTIC plus vaccine: the same vaccination schedule was combined with DTIC (800 mg/mq i.v.) administered one day before each vaccine administration according to the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven diagnosis of melanoma stage II, III, and IV without clinical/radiological evidence of disease
* Age >18 years
* life expectancy of more than 6 months
* ECOG performance status of 0-2
* adequate blood cell counts and kidney-liver function
* use of adequate contraceptive methods
* signed informed consent

Exclusion Criteria:

* concomitant or previous history of malignant disease, except for in situ cervical carcinoma or non melanomatous skin cancer
* severe cardiovascular disease
* clinically active infections and/or significant autoimmune diseases
* concomitant or previous (within 6 weeks) treatment with immunosuppressive drugs
* previous treatments with chemotherapy and/or interferon alpha or beta within 4 weeks and/or radiotherapy within 6 weeks an/or biological therapy within 8 weeks before starting vaccination
* psychiatric illness interfering with patient compliance, pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-09; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Assessment of safety by evaluating local and systemic adverse reactions during the trial. Assessment of the vaccine-specific cellular immune responses | one year

SECONDARY OUTCOMES:
Assessment of relapse-free survival and overall survival calculated from the time of the first chemotherapy/vaccine injection. Evaluation by microarray analysis of the gene expression profiles of patients PBMC 24 h after DTIC administration. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Ferraresi, M.D., Principal Investigator — Regina Elena Cancer Institute; Mario Roselli, M.D., Principal Investigator — University of Rome Tor Vergata; Enrico Proietti, M.D., Study Director — Istituto Superiore di Sanità
Locations (2):
- Italy (2):
  - University Hospital Tor Vergata, Rome
  - Regina Elena Cancer Institute, Rome